CLINICAL TRIAL: NCT03348202
Title: Welfare, Wellbeing and Demographic Change: Understanding Welfare Models
Acronym: EMMY
Status: Completed | Type: Observational
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Åbo Akademi University (Other); SINTEF Health Research (Other); Universidad Autonoma de Madrid (Other); Universita di Verona (Other)
Responsible Party: Sponsor
Other Study IDs: THL/610/6.02.01/2017
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Ageing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Focus Group Participants: Approximately 24 groups (6 per country; Finland, Norway, Spain, Italy) consisting participants aged 80+ recruited from: senior community centres, adult day care centres, nursing homes. Each focus group will comprise from 4 to 8 people. Attempts would be made to create gender-balanced groups.

SUMMARY:
The EMMY Project is an interdisciplinary and mixed methods comparative study on impact of welfare systems on mental wellbeing among the oldest old in Finland, Italy, Norway and Spain, including aspects such as equity, social inclusion, empowerment and participation.

The project will delineate the concept of mental wellbeing at old age by qualitative methods, and will dissect the links between welfare systems and mental wellbeing by quantitative methods. It will support exchange of good policies between EU Member States by performing case studies of existing welfare policies and systems in the four participating countries, and it will develop a new research-based tool for assessing the mental wellbeing impact of welfare policies in old people.

The overarching aim of this interdisciplinary, comparative research project is to improve our knowledge and understanding of how different welfare models and related policies, as well as health and social care service approaches, can benefit from adaptation in order to target mental wellbeing in the oldest-old.

The project will support development of social welfare models in order to incorporate a change of focus from mental disorders to mental wellbeing among old people.

This is important, not only because of the ageing of the European population, but also because of increasing pressures on public finances, within and beyond Europe.

DETAILED DESCRIPTION:
The specific objectives of the EMMY project are:

1. to delineate the concept of mental wellbeing at old age and the links between welfare policies and such wellbeing,
2. to support the exchange of public policies with positive impacts on mental wellbeing at old age through thorough analysis of existing policies and
3. to develop a new research-based tool for assessing the mental wellbeing impact of welfare policies in old people.

Theoretical and instrumental conceptualization of mental wellbeing through participatory focus groups and by a review of instruments used to evaluate wellbeing in the ageing population. A set of gender balanced focus groups with elderly people aged 80+ with different levels of functioning, from each of the participating countries will explore what constitutes wellbeing with suggestions for improvement, building on previous focus group study by Forsman (2013). The nature and intent of the focus group will be explained to potential participants in writing and verbally, and signed consent will be obtained. A manual will guide the focus group procedures, providing open-ended questions for the sessions, and a case report form documenting sociodemographic information. The focus group meetings will be digitally recorded, documented by field notes to pick up features of the session outside the audio transcripts, transcribed verbatim and translated into English. Personal data will be recorded anonymously using identification codes. Data extraction will be performed for qualitative analysis.

Assessment the impact of welfare systems on mental wellbeing in old age, by studying their effect on subjective and personal wellbeing, social inclusion, empowerment, social capital, participation and wider structural determinants of mental health in old age.

Welfare regimes types will be identified using refined and extended versions of the Esping-Andersen typology of welfare regimens (Esping-Andersen 1990, 1999, Ebbinghaus 2012) with quantitative data from existing comparative datasets. Analysis of mental wellbeing among the elderly will be based on data on individual level from European Social Survey (ESS). ESS has been performed in 7 rounds and includes e.g. a core module of subjective wellbeing, social exclusion, religion, national and ethnic identity, as well as rotating modules covering topics relevant to mental wellbeing e.g. personal wellbeing in 2012 round. ESS covers all four partner countries, as opposed to e.g. SHARE or COURAGE data sets. System level variables will be derived from different sources such as ESS Multilevel Data, EU Statistics on Income and Living Conditions (EU-SILC), OECD Social and Welfare Statistics, Social Expenditure Database (SOCX), OECD Health Statistics, Comparative Welfare States Data Set, and Eurobarometers. Analyses will include all European countries in the ESS and respondents above 70 and 80 years (7800 and 2200, respectively). Separation between "young" and "old" elderly as well as using the rest of the adult population as reference group will contribute to interpretation of finding as being age specific or general difference among welfare models. A separation between general and age specific welfare policies will be done. The influence of welfare state regimes and welfare state indicators/dimensions will be performed by use of multilevel regression analysis.

Case studies of welfare models for older people will be produced in each of the participating countries, with a specific emphasis on mental wellbeing. A comparative analysis will produce a qualitative description of promising policies in terms of equity, cost, feasibility and acceptability. The approach will include analyses of the policy processes as well as contextual factors in each country through three actions: a) Case studies, based on comprehensive scoping reviews of existing legislations, initiatives and policies using grey literature; b) Development of a tool to compare existing policies and collect contextual information in each country; c) A qualitative evaluation of existing policies through structured interviews with the main stakeholders.

A scoping review of policies will be performed by focusing on grey literature produced in the four Member States. These will include (as indicative examples) a review of relevant legislations, policies, practices, initiatives, programmes and reports of the Member States governments and agencies and of other national/local relevant organisations. Policies both in health and social domains will be included. In each country partner, local researchers will collate relevant materials in their countries and translate the main non-English documentation. The reviews will result in four case studies to: 1) describe the existing policies, with a specific emphasis on the effectiveness, unintended effects, equity, cost, feasibility and acceptability of the welfare model in relation to mental wellbeing of old people; and 2) identify promising good welfare policies to support mental wellbeing in the oldest-old.

A tool compiled of a battery of checklists/inventories, instruments and indexes will be created, based on a review of existing instruments, for the comparative policy analysis and the description of the contextual factors/system variables. The tool will be based on previous developed instruments for policy analysis (e.g. WHO-AIMS and the REMAST tool, developed by the participant). Data will be collected with the tool using several sources of information: national and international statistics, published national reports and interviews with the main stakeholders and policy makers for welfare systems in each country. A structured deep interview will be created in order to collect stakeholder's views and opinions on existing policies and promising initiatives.

A European tool which raises awareness and understanding of mental wellbeing among the old will be tested and disseminated, enabling stakeholders to identify the impact of a particular policy, service, programme or project may have on it.

Welfare policies have a major impact on mental health determinants. To maximise potential positive impacts, reduce negative impacts on mental health and to reduce mental health inequalities among old people, tools are needed to demonstrate and monitor mental wellbeing impact of policies. Such tools also increase the accountability of policy-makers for mental health impact and will enable a Mental Health in All Policies (MHiAP) approach to promote mental health and wellbeing among old people by initiating and facilitating action within different non health public policy areas. The MHiAP approach can be applied at all administrative levels, ranging from local authorities to the EU level.

The project will develop and disseminate a model for mental health impact assessment of welfare policies, intended for decision makers and stakeholder groups. The tool will target policy decision makers and be freely available in electronic format. Furthermore, the project will suggest a set of indicators to monitor policy impact on mental wellbeing of the oldest old. This will offer policy-makers and stakeholders a tool to compare the situation in different countries and to disentangle the effects of different dimensions as well as single indicators on the overall composite result.

ELIGIBILITY:
Inclusion Criteria:

People aged 80+.

* Cognitive capacity to understand the information sheet and sign the Participant Consent Form and participate in a focus group session according to the moderators' criteria.
* Knowledge of the language of the focus group.
* The individual has been informed of the purpose and rationale of the study, has understood both, and has had all questions answered by the researcher.
* The individual has signed the Participant Consent Form

Exclusion Criteria:

* Individuals who do not have capacity to give informed consent and/or otherwise not able to conform to focus group protocol

Min Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Participants aged 80+ recruited from: senior community centres, adult day care centres, nursing homes. Each focus group will comprise from 4 to 8 people. Attempts would be made to create gender-balanced groups.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Delineate the concept of mental wellbeing at old age by qualitative methods. | 2017-2019
  Qualitative data on mental wellbeing will be collected by representative participatory focus groups in each country (Finland, Norway, Spain Italy).
Investigate the links between welfare systems and mental wellbeing by quantitative methods. | 2017-2019
  Quantitative data will be derived from existing comparative datasets, preferably from datasets that cover all participating countries such as European Social Survey (ESS), European Union Statistics on Income and Living Conditions (EU-SILC), Eurobarometers and from national datasets.

CONTACTS AND LOCATIONS:
Overall Officials: Kristian R Wahlbeck, MD, Principal Investigator — National Institute for Health and Welfare (THL)
Locations (1):
- National Institute for Health and Welfare, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Project website — http://www.emmyproject.eu